CLINICAL TRIAL: NCT03232606
Title: Physical Activity of Asthmatic School Children and Teenagers: Evaluation and Perspectives
Brief Title: Physical Activity of Asthmatic Children
Acronym: Asthmeact
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: University of Lorraine (Other)
Responsible Party: Sponsor
Other Study IDs: N°ID-RCB: 2017-A01483-50
Record Dates: First submitted 2017-06-27; First posted 2017-07-28 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Physical Activity; Asthma; Child Development
MeSH Terms: conditions — Motor Activity; Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Asthmatic children: Asthmatic children aged 6 to 17 year old coming to follow-up at asthma clinic

SUMMARY:
Physical activity is mandatory to the optimal development and health of children. The presence of asthmatic manifestations may influence the comportment of children and its family toward exercise and practice of sports. There no scientific argument to advice a reduction of physical activity in asthmatic children, but previous studies showed that physical activity is reduced in asthmatic children.

The aim of this observational study is to evaluate the existing factors leading to this reduction of physical activity in asthmatic children and their families.

DETAILED DESCRIPTION:
Physical activity is mandatory to the optimal development and health of children. The presence of asthmatic manifestations may influence the behaviour of children and its family with a significant reduction of exercise and practice of sports.

There no scientific argument to advice such a reduction of physical activity in asthmatic children.

The aim of this observational study is to evaluate the existing factors leading to this reduction of physical activity in asthmatic children and their families.

To evaluate the factors explaining this behaviour the investigator design an observational study, based on a questionnaire.

The evaluation of the number of sujets to complete this study is 50 asthmatic children. The whole population will be considered as the same group. This study may be further completed by a comparative and new study including asthmatic and non-asthmatic children.

ELIGIBILITY:
Inclusion Criteria:

* Asthmatic children coming for regular follow-up
* Good control of asthma

Exclusion Criteria:

* Previous pathologies with significant impact on physical activity

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Asthmatic cohort of the asthma clinic of the children hospital
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2017-11-10 (Actual); Study Completion 2017-11-10 (Actual)

PRIMARY OUTCOMES:
Physical activity of children | inclusion visit
  Score

CONTACTS AND LOCATIONS:
Overall Officials: Cyril E SCHWEITZER, MD,PhD, Principal Investigator — University of Lorraine
Locations (1):
- Chru Nancy, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No